CLINICAL TRIAL: NCT00103935
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Examine Safety and Pharmacokinetics of Exenatide Long-Acting Release Administered Weekly in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study Examining Exenatide Long-Acting Release in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2993LAR-104
Record Dates: First submitted 2005-02-17; First posted 2005-02-18 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; long acting release; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A1 (Placebo Comparator): Placebo lead-in followed by placebo equivalent volume to 0.8 mg exenatide LAR
  Interventions: Drug: placebo
- Group A2 (Placebo Comparator): Placebo lead-in followed by placebo equivalent volume to 2.0 mg exenatide LAR
  Interventions: Drug: placebo
- Group B (Experimental): Exenatide lead-in followed by exenatide LAR 0.8 mg weekly
  Interventions: Drug: Exenatide LAR
- Group C (Experimental): Exenatide lead-in followed by exenatide LAR 2.0 mg weekly
  Interventions: Drug: Exenatide LAR

INTERVENTIONS:
Drug: placebo — Subcutaneously injected placebo 0.02 mL twice daily as lead-in followed by once weekly injected amount equivalent to exenatide LAR 0.8 mcg
  Arms: Group A1
Drug: placebo — Subcutaneously injected placebo 0.02 mL twice daily as lead-in followed by once weekly injected amount equivalent to exenatide LAR 2.0 mcg
  Arms: Group A2
Drug: Exenatide LAR — Subcutaneously injected exenatide 5 mcg (0.02 mL) twice daily as lead-in followed by once weekly injected exenatide LAR 0.8 mcg.
  Other Names: Bydureon
  Arms: Group B
Drug: Exenatide LAR — Subcutaneously injected exenatide 5 mcg (0.02 mL) twice daily as lead-in followed by once weekly injected exenatide LAR 2.0 mcg.
  Other Names: Bydureon
  Arms: Group C

SUMMARY:
Exenatide LAR is a long-acting release formulation of exenatide, which is a twice-daily dosage form currently under investigation as a potential treatment for people with type 2 diabetes mellitus. This study will assess the safety, tolerability, and pharmacokinetics of Exenatide LAR administered weekly by subcutaneous injection in people with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes treated with either: *A stable regimen of metformin for a minimum of 3 months, and/or *Diet modification and exercise for a minimum of 3 months.
* Has HbA1c of 7.1% to 11.0%, inclusive.
* Has a body mass index (BMI) of 25 kg/m2 to 45 kg/m2, inclusive.

Exclusion Criteria:

* Received any investigational drug within 3 months prior to screening.
* Is currently treated with any of the following excluded medications: *Thiazolidinediones within 3 months of screening; * Sulfonylureas within 3 months of screening; * Insulin within 1 year of screening.
* Participated previously in an exenatide clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-02; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Assess the safety, tolerability, and pharmacokinetics of exenatide long-acting release (LAR) administered weekly by subcutaneous (SC) injection in subjects with type 2 diabetes (T2DM) | Time intervals: 0 min to 12 hours on Day 1 for a duration of 12 hours, from Day 1; 0 mininutes to Week 1 for a duration of 168 hours, and from Week 14 to Week 15 for a duration of 168 hours

SECONDARY OUTCOMES:
Examine the effect on various pharmacodynamic parameters of exenatide LAR administered weekly by subcutaneous injection in subjects with Type 2 Diabetes Mellitus | Various time intervals from Day 1 to Week 15
Change in HbA1c (glycosylated hemoglobin) from Baseline to Week 15 and to each intermediate visit where applicable, and to study termination (Week 27). | Day -3, Day 1, Weeks 1, 2, 4, 5, 7, 8, 10, 11, 13, 14, 15, 16, 17, 18, 19, 27
  Change in HbA1c from baseline Visit 3 (Day -3) to Visit 25 (Week 15) and to each intermediate visit where applicable, and to study termination.
Change in fasting glucose concentrations from Baseline to Week 15 and to each intermediate visit where applicable, and to study termination (Week 27) | Day -3, Day 1, Weeks 1, 2, 4, 5, 7, 8, 10, 11, 13, 14, 15, 16, 17, 18, 19, 27
  Change in fasting glucose concentrations from baseline Visit 3 (Day -3) to Visit 25 (Week 15) and to each intermediate visit where applicable, and to study termination
Change in body weight from Baseline to Week 15 and to each intermediate visit where applicable, and to study termination (Week 27) | Day -3, Day 1, Weeks 1, 2, 4, 5, 7, 8, 10, 11, 13, 14, 15, 16, 17, 18, 19, 27
  Change in body weight (kg) from baseline Visit 3 (Day -3) to Visit 25 (Week 15) and to each intermediate visit where applicable, and to study termination
Change in seven-point glucose concentrations from Baseline to Week 14 and Week 15 | Baseline, 3 days between Day -7 and Day -3, and 3 days between Week 14 and Week 15
  Change in seven-point glucose concentrations from baseline (collected on 3 days between Visit 2 [Day -7] and Visit 3 [Day -3]) to Visit 25 (collected on 3 days between Visit 20 [Week 14] and Visit 25 [Week 15])

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (7):
- United States (7):
  - Research Site, Walnut Creek, California
  - Research Site, Honolulu, Hawaii
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Portland, Oregon
  - Research Site, San Antonio, Texas
  - Research Site, Olympia, Washington

REFERENCES:
- [Derived] Fineman M, Flanagan S, Taylor K, Aisporna M, Shen LZ, Mace KF, Walsh B, Diamant M, Cirincione B, Kothare P, Li WI, MacConell L. Pharmacokinetics and pharmacodynamics of exenatide extended-release after single and multiple dosing. Clin Pharmacokinet. 2011 Jan;50(1):65-74. doi: 10.2165/11585880-000000000-00000. PMID 21142268